CLINICAL TRIAL: NCT00441922
Title: A Multicenter Randomized Phase II Study of Docetaxel Versus Vinorelbine as First-Line Treatment in Elderly Patients With Advanced Non-Small-Cell Lung Cancer (NSCLC)
Brief Title: Trial of Docetaxel Versus Vinorelbine as 1st Line Treatment in Elderly Patients With Non-Small-Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: L.Vamvakas, Hellenic Oncology Research Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/03.07
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Cancer; Elderly; Chemotherapy; Docetaxel; Vinorelbine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Docetaxel; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): D
  Interventions: Drug: Docetaxel
- 2 (Experimental): V
  Interventions: Drug: Vinorelbine

INTERVENTIONS:
Drug: Docetaxel — Docetaxel at the dose of 38 mg/m2 IV on days 1 and 8 every 3 weeks for 6 consecutive cycles
  Other Names: Taxotere
  Arms: 1
Drug: Vinorelbine — Vinorelbine at the dose of 25 mg/m2 IV on days 1 and 8 every 3 weeks for 6 consecutive cycles
  Other Names: Navelbine
  Arms: 2

SUMMARY:
This trial will compare the efficacy of docetaxel versus vinorelbine as first-line treatment in elderly patients with advanced NSCLC.

DETAILED DESCRIPTION:
Docetaxel and vinorelbine are well known active agents in the treatment of NSCLC. The standard treatment of elderly patients with advanced NSCLC is monotherapy with a third generation agent. The role of comprehensive geriatric assessment in treatment efficacy and tolerance is an area of investigation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically- confirmed Non-Small-Cell Lung Cancer
* Stage IIIB/IV
* No prior chemotherapy
* Existence of two-dimensional measurable disease. The measurable disease should not have been irradiated
* Life expectancy of more than 3 months
* Age ≥ 65 years
* Performance status (WHO) ≤ 3
* Adequate bone marrow function (absolute neutrophil count > 1000/mm^3, platelet count > 100000/mm^3, Hemoglobin > 9 gr/mm^3)
* Adequate liver (bilirubin < 1.5 times upper limit of normal and SGOT/SGPT < 2 times upper limit of normal), and renal function (creatinine < 2 mg/dl)
* Informed consent

Exclusion Criteria:

* Psychiatric illness or social situation that would preclude study compliance.
* Other concurrent uncontrolled illness
* Other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No absence or irradiated and stable central nervous system metastatic disease.
* No presence of a reliable care giver
* Other concurrent investigational agents

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2003-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Overall survival between the two treatment arms | 1 year

SECONDARY OUTCOMES:
Time to disease progression | 1 year
Toxicity profile | During the time of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Lampros Vamvakas, MD, Principal Investigator — University Hospital of Crete, Department of Medical Oncology
Locations (10):
- Greece (10):
  - University General Hospital of Alexandroupolis, Department of Medical Oncology, Alexandroupoli
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - IASO General Hospital of Athens, 1st Department of Medical Oncology, Athens
  - Laikon General Hospital, Medical Oncology Unit, Propedeutic Department of Internal Medicine, Athens
  - Sismanogleio General Hospital, 1st, 2nd Department of Pulmonary Diseases, Athens
  - Sotiria General Hospital, 1st, 3rd, 8th Department of Pulmonary Diseases, Athens
  - State General Hospital of Larissa, Department of Medical Oncology, Larissa
  - Metaxa's Anticancer Hospital of Piraeus, 1st Department of Medical Oncology, Piraeus
  - Theagenion Anticancer Hospital of Thessaloniki, Thessaloniki